CLINICAL TRIAL: NCT02297386
Title: Phase I Trial Of [18F] Dihydro-testosterone Pet and MR Imaging In Patients With Localized Prostate Cancer
Brief Title: [18F] Dihydro-testosterone Pet and MR Imaging In Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-185
Record Dates: First submitted 2014-11-18; First posted 2014-11-21 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer; Localized Prostate Cancer
Keywords: [18F] Dihydro-testosterone; PET Scan; MRI; 14-185
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron-Emission Tomography; Blood Specimen Collection

ARMS (1):
- [18F] DIHYDRO-TESTOSTERONE PET (Experimental): The diagnostic intervention of this study is the use of FDHT PET in localized prostate cancer. Patients will undergo a 30 minute dynamic scan of the pelvis followed by a whole body scan of approximately 30-minutes duration. The dynamic scan will be optional, but strongly encouraged. PET scanning will preferably be done on the GE Discovery STE PET/CT scanner or the equivalent generation of scanner. The PET scans are routinely "quantitative," that is corrected for attenuation and scatter and adjusted for system sensitivity and providing parametric images in terms of standardized uptake values (SUV) (= μCi found/gm tissue / μCi injected/gm body mass).
  Interventions: Drug: [18F] DIHYDRO-TESTOSTERONE; Device: PET scan; Device: MRI; Other: Blood draw

INTERVENTIONS:
Drug: [18F] DIHYDRO-TESTOSTERONE
Device: PET scan
Device: MRI
Other: Blood draw

SUMMARY:
The purpose of this study is to test the ability of a new PET scan radiotracer, called FDHT (stands for [18F] Dihydro-Testosterone), to better find and monitor prostate cancer. Radiotracers are a type of drug that carries small amounts of radioactivity that can be seen by the PET scanner. FDHT is a radiotracer that looks for a protein which is present in almost all prostate cancer cells. The investigators want to find out if we can find and monitor changes in cancer using a FDHT PET scan.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 21 years or older and below 80 years of age.
* Signed written informed consent and willingness to comply with protocol requirements.
* Histologically confirmed diagnosis of prostate cancer.
* Staging imaging workup including a baseline MRI of the prostate and pelvis performed at MSKCC.
* Baseline imaging to rule out distant metastatic disease (99mTc bone scan, NaF PET, total body MRI, or CT chest/abdomen/pelvis)
* Karnofsky performance status ≥ 70
* Clinical criteria required to be eligible:

  a. One of the following i.Pre-treatment PSA ≥10 ng/dL, OR ii. Clinical T-stage assessed by digital rectal exam of ≥T2a, OR ii . Radiographic ≥T3a on MRI, OR iv. Gleason score of ≥3+4=7 c. Visible intraprostatic tumor foci ≥1 cm in largest dimension on T2-weighted images based on initial pre-treatment MRI
* Physician recommendation of ADT.

Exclusion Criteria:

* Metastatic disease on standard staging imaging (beyond regional lymph node involvement).

  o Absence of metastatic disease (beyond regional lymph node involvement) as defined by a negative bone scan, NaF PET, CT chest/abdomen/pelvis, or total body MRI.
* Prior treatment of the prostate gland for malignant conditions (surgery, cryotherapy, radiotherapy, or photodynamic therapy).
* Physician prescription of androgen receptor antagonist therapy (examples: bicalutamide, flutamide, or enzalutamide) during time of protocol scans.

  o Note: ADT consists of chemical castration (i.e. degarelix) to remove endogenous DHT. Androgen receptor antagonists will bind to the androgen receptor and inhibit FDHT from binding.
* Patients receiving testosterone supplementation .
* Any contraindication to baseline MRI based on departmental MR questionnaire, or inability to cooperate for an MRI scan.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to FDHT.
* Hepatic laboratory values:

  1. Bilirubin >1.5 x ULN (institutional upper limits of normal)
  2. AST/ALT >2.5 x ULN
  3. Albumin <2 g/dL
* Creatinine >2.5 mg/dL
* Calcium >11 mg/dL
* Other serious illness(es) which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study.

Ages: 21 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
increase in standardize uptake values (SUV) between the second and third FDHT scans | 1 year
  Enrolling 15 patients will provide 80% power to detect a 33% increase in the mean uptake (from 6 to 8) between the 2nd and the 3rd scans.

SECONDARY OUTCOMES:
correlate AR expression to FDHT uptake | 1 year
  involves collecting formalin fixed paraffin embedded tissue from pre-treatment biopsy specimens to correlate androgen receptor (AR) expression to FDHT uptake. AR expression will be measured using RNA-seq and correlated with FDHT SUV values separately for each scan using Spearman's rank correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Osborne, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/